CLINICAL TRIAL: NCT07341698
Title: Prehabilitation for Patients Diagnosed With Blood Cancer and Treated With Alloge-neic Hematopoietic Stem Cell Transplantation - a National Randomized Controlled Trial
Brief Title: Prehabilitation for Patients Diagnosed With Blood Cancer and Treated With Al-logeneic Hematopoietic Stem Cell Transplantation
Acronym: PrepAllo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Jan Christensen, Senior Researcher and Head of Research, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-25053677; MS25-01447 (Other Grant/Funding Number: Danish Cancer Society)
Record Dates: First submitted 2025-12-10; First posted 2026-01-14 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Allogeneic Hematopoietic Stem Cell Transplantation Recipient
Keywords: Prehabilitation; Exercise; resistance training; nutritional support
MeSH Terms: conditions — Motor Activity | interventions — Resistance Training; Exercise; Preoperative Exercise; Nutritional Support; Nutrition Assessment; Nutritional Status; Hematopoietic Stem Cell Transplantation

STUDY DESIGN:
Intervention Model Description: This study is a multicenter RCT. Based on a 1:1 randomization ratio, participants will be allo-cated to either usual care or usual care plus the prehabilitation intervention.
Who Masked: Outcomes Assessor
Masking Description: Outcomes Assessor and statistician will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (Active Comparator): The usual care group will receive standard care, including physio- and occupational therapy if admitted to the hospital, and potentially referral to rehabilitation in the municipality three months after transplantation.
  Interventions: Procedure: Usual care
- Usual care plus the prehabilitation intervention (Experimental): The prehabilitation group will in addition to usual care receive supervised individually tailored resistance training and optimized nutritional support
  Interventions: Other: Resistance training; Dietary Supplement: Nutritional Support; Procedure: Usual care

INTERVENTIONS:
Other: Resistance training — Structured and supervised, group-based, resistance training 3x per week (individually tailored to the individual's capabilities)
  Other Names: Exercise; Prehabilitation
  Arms: Usual care plus the prehabilitation intervention
Dietary Supplement: Nutritional Support — Optimized dietary counseling and supplementation to optimize nutritional intake
  Other Names: Prehabilitation; dietary counseling; nutrition
  Arms: Usual care plus the prehabilitation intervention
Procedure: Usual care — Usual care is the standard care before allogeneic hematopoietic stem cell transplantation
  Other Names: HSCT; allogeneic hematopoietic stem cell transplantation; hematopoietic stem cell transplantation

SUMMARY:
Seventy-five percent of patients treated with hematopoietic stem cell transplants survive one-year post-transplantation. However, this intensive treatment is associated with prolonged hospitalizations and significant deconditioning. Pathophysiological changes in skeletal muscle mass and function have notable implications for disease progression and long-term prognosis. Patients frequently report substantial rehabilitation needs, though these needs are highly individualized and fluctuate over time, with musculoskeletal dysfunction and fa-tigue being the most common barriers to prehabilitation. Furthermore, at least 35% of cancer patients are found to have inadequate daily protein intake, which may hinder improve-ments in physical performance through prehabilitation. Several recent studies have demonstrated the safety and feasibility of exercise-based prehabilitation interventions during the pre-transplant period. However, no full-scale randomized controlled trial (RCT) has been conducted to date.

DETAILED DESCRIPTION:
Evaluate the effectiveness of an individualized prehabilitation intervention in addition to usual care, compared to usual care alone on HRQoL, and secondary outcomes hospitalization, muscle mass and muscle function.

ELIGIBILITY:
Inclusion Criteria:

Adult patients >18 years will be eligible for inclusion if they are scheduled for a allo-HSCT with at least four weeks before their scheduled transplantation date.

Exclusion Criteria:

* pregnancy
* physical or mental disabilities precluding test of muscle function
* inability to read and understand Danish or English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2026-01-12 (Actual); Primary Completion 2028-01-12 (Estimated); Study Completion 2032-10-12 (Estimated)

PRIMARY OUTCOMES:
Health-Related Quality of Life using European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Core questionnaires with 30 questions (EORTC QLQ C-30) | From enrollment to 90 days post-transplantation
  HRQoL measured using EORCT-C30v3.0. Scores are from 0 to 100 with lower scores meaning poorer quality of life and high scores meaning better overall quality of life.

SECONDARY OUTCOMES:
Hospitalization | From enrollment to 90 days post-transplantation
  Days of hospitalization
Appendicular lean mass | From enrollment to 90 days post-transplantation
  Measured using dual-energy X-ray absorptiometry (DXA)
Appendicular Lean Mass Index | From enrollment to 90 days post-transplantation
  To account for body size, ALM is divided by height squared
Hand grip strength | From enrollment to 90 days post-transplantation.
  Using a handheld electronical dynamometer
Lower limb strength | From enrollment to 90 days post-transplantation.
  5-repetition Sit-to-stand Test
Lower limb strength and endurance | From enrollment to 90 days post-transplantation.
  30-second Sit-to-stand Test
Leg Extensor Power | From enrollment to 90 days post-transplantation
  Measured using a Nottingham Power Rig,

OTHER OUTCOMES:
Habitual gait speed | From enrollment to 90 days post transplantation
  10-Meter walk test: Time to walk 10 meter distance at a preferred speed
Physical activity monitoring monitored with the use og SENS motion wearable activity sensors. Outcome will be reported in metabolic equivalents (METS) | From enrollment to 90 days post-transplantation
  Moderate to Vigorous Physical Activity (MVPA) will be measured with algorithms from the use of SENS motion wearables
Physical activity monitoring | From enrollment to 90 days post-transplantation
  Daily steps
Self reported physical activity | From enrollment to 90 days post-transplantation
  International Physical Activity Questionnaire short form (IPAQ-sf)
Karnofsky Performance Status | From enrollment to 90 days after transplantation
  Changes in Karnofsky Performance Status. Minimum value is 0 and maximum value is 100. A score of 100 equals normal function in performing daily activities while a score of 0 is equal to death. Thus, the lower scores the poorer performance of daily activities.
Symptoms of anxiety using Hospital Anxiety and Depression Scale (HADS) | From enrollment to 90 days post-transplantation
  Symptoms of anxiety measured using HADS. The item is separated in two parts. One is scoring anxiety level and one is scoring depression level. The minimum value is 0 while the maximum for each scale is 21 for each scale (21 for anxiety and 21 for depression). The higher score the more severe symptoms of either anxiety or depression. Scores above 11 in each category is considered to be moderate to severe symptoms with action needed to be taken on the condition.
Symptoms of depression using Hospital Anxiety and Depression Scale (HADS) | From enrollment to 90 days post-transplantation
  Symptoms of depression measured using HADS. Symptoms of anxiety measured using HADS. The item is separated in two parts. One is scoring anxiety level and one is scoring depression level. The minimum value is 0 while the maximum for each scale is 21 for each scale (21 for anxiety and 21 for depression). The higher score the more severe symptoms of either anxiety or depression. Scores above 11 in each category is considered to be moderate to severe symptoms with action needed to be taken on the condition.
Health literacy mesured using the Health Literacy Questionnaire (HLQ). | From enrollment to 90 days post-transplantation
  Health literacy was assessed using the Health Literacy Questionnaire (HLQ). The HLQ comprises nine independent scales scored as the mean of their constituent items. Scales 1-5 are scored from 1 to 4, and scales 6-9 from 1 to 5, with higher scores indicating better health literacy.
Days of hospitalization | From enrollment to 90 days and 1, 3 and 5 years after transplantation
  Days of hospitalization
Survival | 1, 3 and 5 years after transplantation
  All-course survival with-out progression or relapse
Interviews | Participants will be asked to participate in interviews at time for recruitment (6-8 weeks before transplantation), at end of interventionperiod (day -7 to 0 before transplantation) and after last follow-up tests at day +90 after transplantation.
  Participants will be asked to participate in interviews during the study period
Complete remission | at day +90 and 1,3 and 5 years after transplantation
  Complete remission objective measured and evaluated by responsible physician. Complete remission is defined as full donor dhimerism if >95 % of bone marrow cells measured from chimerism is from donor.
Cancer Progression | At 1, 3 and 5 years after transplantation
  Progression of the underlying hematologic malignancy will be defined as objective worsening of disease burden after transplantation among patients who have not achieved complete remission after HSCT
Cancer recurrence | 1,3 and 5 years after transplantation
  Recurrence (relapse) will be defined as reappearance of the original hematologic malignancy in a patient who has previously achieved complete remission after HSCT
Exercise habits | 1,3 and 5 years after transplantation
  Exercise habits rapported by International Physical Activity Questionnaire (IPAQ)
Secondary malignancy | At 1, 3 and 5 years after transplantation
  Secondary malignancy will be defined as the occurrence of any new hematologic or solid malignant disease after HSCT that is genetically or clinically distinct from the primary malignancy for which the transplant was performed.
Engraftment | From enrollment to 90 days after transplantation
  Time from transplantation to first of three following days with absolute neutrophiles >0,5 x10^9 /L
Transfusion need | From day 0 to day 90
  Days after transplantation with being independent of bloodtransfusions
Acute GvHD | Development of > grade 2 Acute GvHD from day 0 to day 90
  Development of Acute GvHD

CONTACTS AND LOCATIONS:
Locations (1):
- Copenhagen University Hospital - Rigshospitalet, Copenhagen, Denmark, Denmark

IPD SHARING:
Plan to Share IPD: Yes
The investigators have agree to make data and materials supporting the results and analyses available upon reasonable request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code